CLINICAL TRIAL: NCT02284646
Title: Assessment of the Efficacy of a Physical Training Program in Patients With Ankylosing Spondylitis
Brief Title: Physical Training Program in Ankylosing Spondylitis
Acronym: PEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 7027 08
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2020-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Physical training program
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized physical training (Experimental): 9-week personalized physical training program (ergometric bicycle)
  Interventions: Other: Personalized physical training program
- Information about physical activity (No Intervention): 2 sessions of information on physical activity

INTERVENTIONS:
Other: Personalized physical training program — 9-week personalized physical training program (ergometric bicycle)
  Arms: Personalized physical training

SUMMARY:
Purpose: to assess the efficacy of a physical training program in patients with ankylosing spondylitis (AS) in a randomized controlled study

DETAILED DESCRIPTION:
AS is a chronic inflammatory rheumatic disorder affecting spine, peripheral joints and entheses. Patients undergo pain, stiffness and reduced mobility of spine and joints. Patients experience limitations in physical activities and reduced quality of life. Some uncontrolled studies reported benefits of physical activity in patients with AS.

The aim of the present study is to assess the efficacy of a physical training program in patients with AS.

Patients will be randomized in two parallel arms: program of personalized physical training (intervention group [PEPc]) or program of information about physical activity (control group [PIAP]).

Patients will be evaluated at 12 and 24 weeks on activity, functional and metrological scores (ASAS 20, ASAS 5/6, ASDAS, BASDAI, BASFI, BASMI); biological inflammation (CRP); NSAID use and pain VAS.

Primary outcome: percentage of patients reaching an ASAS 20 response at 12 weeks.

Secondary outcomes: ASAS 20 at 24 weeks, ASAS5/6, ASDAS, BASDAI, BASFI, BASMI, CRP, NSAID use and pain VAS at 12 and 24 weeks.

Statistical analysis: comparison of the percentage of patients reaching an ASAS 20 response at 12 weeks in each arm using a Fisher's exact test (main outcome).

ELIGIBILITY:
Inclusion Criteria:

* Patients with AS according to ASAS criteria,
* treated or not with NSAID,
* synthetic DMARD or anti-TNF agent.

Exclusion Criteria:

* Contraindications to physical training program (e.g. cardiac failure, pregnancy, painful arthroplasty or lower limbs damaged joint).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching an ASAS 20 response | Week 12

SECONDARY OUTCOMES:
Percentage of patients reaching an ASAS 20 response | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud constantin, MD, PHD, Principal Investigator — UH Toulouse
Locations (1):
- University Hospital, Toulouse, France

REFERENCES:
- [Result] Pecourneau V, Degboe Y, Barnetche T, Cantagrel A, Constantin A, Ruyssen-Witrand A. Effectiveness of Exercise Programs in Ankylosing Spondylitis: A Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2018 Feb;99(2):383-389.e1. doi: 10.1016/j.apmr.2017.07.015. Epub 2017 Aug 30. PMID 28860095